CLINICAL TRIAL: NCT04933708
Title: The Effect of a Labor Podcast Intervention on Patient Satisfaction and Postpartum Depression in Nulliparous Women
Brief Title: LaPPS: Labor Podcast for Patient Satisfaction
Acronym: LaPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Fei Cai, MD, Professor of Obstetrics and Gynecology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 848622
Record Dates: First submitted 2021-06-13; First posted 2021-06-22 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Labor Onset and Length Abnormalities; Pregnancy Related
Keywords: Nulliparity; Podcast; Labor

STUDY DESIGN:
Intervention Model Description: Pregnant patients between 28w0d - 36w0d will be randomized to one of the following study arms upon enrollment. Patients will be approached after 20 weeks for consent and randomized after they reach 28 weeks. The study will be done in an intent-to-treat fashion. Due to the nature of the study, blinding will not be possible.
  Study Arms
  1. Labor Podcast Group
  2. Usual Teaching
Who Masked: Care Provider
Masking Description: Those that provide care for patients on the labor floor will not know if they have had access to labor podcasts or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor Podcast Group (Experimental): 1) Labor Podcast Group - Women randomized to this arm will receive access to a link to download six HUP physician created labor podcasts in addition to usual care during labor, delivery, and postpartum
  o Podcast topics: Labor Anesthesia, Induction of Labor, Second Stage of Labor, Reasons for Cesarean Section, Postpartum Recovery, Complications of Labor and Birth
  * LAS-10 and Birth Satisfaction survey - Women will be sent these surveys on postpartum day 2 via method they indicated they desire (either email or text message)
  * EPDS - Women will receive this survey on postpartum day 7 via method they desire
  Interventions: Behavioral: Labor Podcast
- Usual Care (No Intervention): 2. Usual care Women randomized to this arm will receive usual care during labor, delivery, and postpartum with the following exceptions:
  * LAS-10 and Birth Satisfaction survey Women will be sent these surveys on postpartum day 2 via method they indicated they desire (either email or text message)
  * EPDS Women will receive this survey on postpartum day 7 via method they desire

INTERVENTIONS:
Behavioral: Labor Podcast — Listening to podcasts.
  Topics include:
  Labor Anesthesia, Induction of Labor, Second Stage of Labor, Reasons for Cesarean Section, Postpartum Recovery, Complications of Labor and Birth
  Arms: Labor Podcast Group

SUMMARY:
Patients will be enrolled at 28w0d-36w0d. Randomized to one of two arms:

1. Labor podcasts - Seven labor podcasts that can be downloaded for any podcast app
2. Usual care

DETAILED DESCRIPTION:
Objectives Overall objectives To assess the effect of listening to physician-created podcasts of common labor topics on patient satisfaction and perception of their birth experience Primary outcome variable(s) Patient satisfaction as measured by LAS + 2 satisfaction questions Secondary outcome variable(s) Edinburgh Postpartum Depression Scale (EPDS) scores Logistic regression for multivariate analysis with regards to demographics and other birth outcomes

Background Recently, podcasts have been used for both undergraduate and graduate medical education, with studies showing that they are feasible, acceptable, and effective. Learners appear to enjoy podcast learning because they increased efficiency by allowing listeners to multitask, made listeners keep up to date with medical literature, and increased overall knowledge. However, podcast learning has not been as widespread for patient education. There have been some studies that showed that podcast patient education is feasible, and one small study showed increased knowledge scores after listening to podcasts.

To our knowledge, podcast learning has never been studied in the obstetric population. Labor and delivery is usually a time that is fraught with questions from first time mothers, and more education may increase these women's perception of control and satisfaction overall with birth and the postpartum period. The Labor Agentry Scale (LAS)-10 is a validated instrument measuring expectancies and experiences of personal control during childbirth. The Edinburgh Postnatal Depression Scale (EPDS) is also a validated scale that measures levels of postpartum depression that is commonly used at our institution both immediately postpartum and at the postpartum visit 4-6 weeks after delivery.

Study Design Design Pregnant patients between 28w0d - 36w0d will be randomized to one of the following study arms upon enrollment. Patients will be approached after 20 weeks for consent and randomized after they reach 28 weeks. The study will be done in an intent-to-treat fashion. Due to the nature of the study, blinding will not be possible.

Study Arms 1) Labor Podcast Group - Women randomized to this arm will receive access to a link to download seven HUP physician created labor podcasts in addition to usual care during labor, delivery, and postpartum

o Podcast topics: Labor Anesthesia, Induction of Labor, Second Stage of Labor, Reasons for Cesarean Section, Postpartum Recovery, Complications of Labor and Birth, Normal Labor

* LAS-10 and Birth Satisfaction survey - Women will be sent these surveys on postpartum day 2 via method they indicated they desire (either email or text message)
* EPDS - Women will receive this survey on postpartum day 7 via method they desire

  2. Usual care Women randomized to this arm will receive usual care during labor, delivery, and postpartum with the following exceptions:
* LAS-10 and Birth Satisfaction survey Women will be sent these surveys on postpartum day 2 via method they indicated they desire (either email or text message)
* EPDS Women will receive this survey on postpartum day 7 via method they desire

Study duration Estimated length of time to enroll all subjects and complete the study Length of a subject's participation time in study Project date of the proposed study

Estimated length of time to enroll all subjects and complete study:

Based on previous studies using the LAS-10, average score ranged between 45-53/70, with standard deviations ranging from 6-12. Therefore, we would estimate that the LAS score in the usual care group to be approximately 50. To be able to detect an effect size of 4, with a standard deviation of 9, and to achieve a power of 0.8 and alpha of 0.05, we would need a sample size of approximately 79 subjects per group. Calculating for a 20% loss to follow-up rate, we would anticipate recruiting 95 subjects per group.

Our city has an average of 16% preterm birth rate. Our hospital averages 1400 nulliparous deliveries/year. We would conservatively estimate approaching 50% of these women in the prenatal period for enrollment. If we assume a 75% consent rate for the RCT, which is standard for our center, we anticipate enrolling 30-36 women per month in our study. We would therefore anticipate it taking 6 months before we reach our target sample size.

We would then require an additional 6 months to compile and analyze the data.

Length of subject's participation:

Women will be followed from time of consent until 7 days postpartum Women will be followed from time of consent until 7 days postpartum.

Project date of the proposed study:

Proposed to start April 2021 for recruitment and enrollment. We anticipate enrolling all patients by end of September 2021. We would likely be able to conclude the study by April 2022.

Resources necessary for human research protection Subjects will be recruited from looking at antepartum clinic charts and messaged via MPM once they are deemed eligible. This can be one by Dr. Cai and Dr. Srinivas. Both will be trained in the study protocol prior to enrolling subjects.

The research staff will also distribute information regarding the study to the aforementioned prenatal clinics so that written information can be handed out by providers to patients. This will allow for patients to be aware of the study. However, only study personnel will be able to consent and enroll patients.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Singleton pregnancy
* English-speaking
* Age 18-50
* Own a smart phone or device capable of downloading podcasts
* Reached at least 36w0d of gestation
* Willing and able to sign consent form

Exclusion Criteria:

* Planned cesarean delivery
* Complication in pregnancy including:

  * Placenta accrete spectrum
  * Vasa previa
  * Intrauterine fetal demise
  * Known major fetal anomaly
* Delivery planned at location other than the Hospital of the University of Pennsylvania

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sindhu Srinivas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SC, Huang H, Minard CG, Schackman J, Rajagopalan S. The use of podcast videos for airway skills. Clin Teach. 2019 Dec;16(6):585-588. doi: 10.1111/tct.12984. Epub 2018 Dec 27. PMID 30592144
- [Background] Cai F, Burns RN, Kelly B, Hampton BS. CREOGs Over Coffee: Feasibility of an Ob-Gyn Medical Education Podcast by Residents. J Grad Med Educ. 2020 Jun;12(3):340-343. doi: 10.4300/JGME-D-19-00644.1. PMID 32595856
- [Background] Young B, Pouw A, Redfern A, Cai F, Chow J. Eyes for Ears-A Medical Education Podcast Feasibility Study. J Surg Educ. 2021 Jan-Feb;78(1):342-345. doi: 10.1016/j.jsurg.2020.06.041. Epub 2020 Jul 21. PMID 32709568
- [Background] Malecki SL, Quinn KL, Zilbert N, Razak F, Ginsburg S, Verma AA, Melvin L. Understanding the Use and Perceived Impact of a Medical Podcast: Qualitative Study. JMIR Med Educ. 2019 Sep 19;5(2):e12901. doi: 10.2196/12901. PMID 31538949
- [Background] Chin A, Helman A, Chan TM. Podcast Use in Undergraduate Medical Education. Cureus. 2017 Dec 9;9(12):e1930. doi: 10.7759/cureus.1930. PMID 29464137
- [Derived] Cai F, McCabe M, Srinivas SK. A randomized trial assessing the impact of educational podcasts on personal control and satisfaction during childbirth. Am J Obstet Gynecol. 2023 May;228(5):592.e1-592.e10. doi: 10.1016/j.ajog.2023.01.021. Epub 2023 Feb 13. PMID 36791987

RESULTS

PARTICIPANT FLOW:
Groups:
- Labor Podcast Group: 1) Labor Podcast Group - Women randomized to this arm will receive access to a link to download six HUP physician created labor podcasts in addition to usual care during labor, delivery, and postpartum
  o Podcast topics: Labor Anesthesia, Induction of Labor, Second Stage of Labor, Reasons for Cesarean Section, Postpartum Recovery, Complications of Labor and Birth
  * LAS-10 and Birth Satisfaction survey - Women will be sent these surveys on postpartum day 2 via method they indicated they desire (either email or text message)
  * EPDS - Women will receive this survey on postpartum day 7 via method they desire
  Labor Podcast: Listening to podcasts.
  Topics include:
  Labor Anesthesia, Induction of Labor, Second Stage of Labor, Reasons for Cesarean Section, Postpartum Recovery, Complications of Labor and Birth
Period: Overall Study
Arm/Group | Labor Podcast Group | Usual Care
Started | 101 | 100
Completed | 78 | 75
Not Completed | 23 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Labor Podcast Group | Usual Care | Total
Number analyzed (Participants) | 78 | 75 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 75 | 153
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.26) | 29.3 (6.08) | 30 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 24 | 47
  White | 38 | 35 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 78 | 75 | 153

OUTCOME MEASURES:

1. Primary Outcome: Labor Agentry Scale
Description: Subjects will complete the labor agentry scale after delivery. Score on labor agentry scale will be compared between groups. Score range: 10-70. Higher scores indicate more agentry, which we consider to be better for this study.
Time Frame: 2 days after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Labor Podcast Group | Usual Care
Number analyzed (Participants) | 78 | 75
score on a scale | 57 [50 to 63] | 54 [47 to 62]

2. Secondary Outcome: Birth Satisfaction
Description: Subjects will also complete a birth satisfaction survey after delivery. Score on birth satisfaction will be compared between two groups. Score range: 3 - 21. Higher scores indicate higher satisfaction.
Time Frame: 2 days after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Labor Podcast Group | Usual Care
Number analyzed (Participants) | 78 | 75
score on a scale | 20 [18 to 21] | 18 [16 to 21]

3. Secondary Outcome: Edinburgh Postpartum Depression Scale
Description: Subjects will complete the EPDS 7 days postpartum. Scores will be compared between the two groups. Score range: 0-30. Higher scores indicate more risk of depression
Time Frame: 7 days postpartum
Population: Subjects are same as previously described
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Labor Podcast Group | Usual Care
Number analyzed (Participants) | 78 | 75
score on a scale | 4 [1 to 5] | 3 [1 to 7]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed for this trial.
Arm/Group | Labor Podcast Group | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04933708/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04933708/ICF_001.pdf